CLINICAL TRIAL: NCT02761551
Title: Centralized IIS-based Reminder/Recall to Increase Childhood Influenza Vaccination Rates: Colorado
Brief Title: Centralized IIS-based Reminder/Recall to Increase Childhood Influenza Vaccination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-0570
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Reminder Systems; Influenza Vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual Care (No Intervention): Patients in this group will not receive any reminders for influenza vaccine.
- 1 notice (Experimental): Patients in this group will receive one reminder for influenza vaccine across the 2016 influenza season.
  Interventions: Behavioral: Reminder notifications via autodialer
- 2 notices (Experimental): Patients in this group will receive up to two reminders for influenza vaccine across the 2016 season.
  Interventions: Behavioral: Reminder notifications via autodialer
- 3 notices (Experimental): Patients in this group will receive up to three reminders for influenza vaccine across the 2016 season.
  Interventions: Behavioral: Reminder notifications via autodialer

INTERVENTIONS:
Behavioral: Reminder notifications via autodialer
  Arms: 1 notice; 2 notices; 3 notices

SUMMARY:
Despite U.S. guidelines for influenza vaccination of all children starting at age 6 months, only about half of children are vaccinated annually leading to substantial influenza disease in children and spread of disease to adults. A major barrier is that families are not reminded about the need for their children to receive influenza vaccination. The investigators will evaluate the impact of patient reminder/recall (R/R) performed by state immunization information systems to improve influenza vaccination rates by using three clinical trials in two states. The investigators will assess effectiveness and cost-effectiveness of phone reminder/recall on improving influenza vaccination rates. The investigators will disseminate the state immunization information system based reminder/recall system to all states for use for both seasonal and pandemic influenza vaccinations with the goal of lowering influenza morbidity.

DETAILED DESCRIPTION:
Annual epidemics of seasonal influenza cause substantial morbidity and mortality in the U.S. with high rates of hospitalizations, emergency department and outpatient visits, and medical costs. Children experience significant morbidity from influenza, and also play a critical role in spreading infection to adults. Since 2010, the Advisory Committee on Immunization Practices (ACIP) has recommended influenza vaccination for all children >6 months of age. However, vaccination rates remain very low-- only 56% of children 2-17 years are vaccinated. Low rates are a concern for both seasonal influenza and in preparation for pandemic influenza. One of the nationally recommended strategies for raising childhood influenza vaccination rates is to use parent reminder/recall (R/R) by phone or mail, which can raise rates by up to 20 percentage points. However, less than 16% of primary care practices use R/R despite many studies showing its effectiveness.

Statewide immunization information systems (IISs) now exist in all states to track childhood vaccinations, but they have not been used for R/R for influenza vaccine because of the lack of evidence for its effectiveness and lack of a template for IIS-based R/R. The investigators have united two leading immunization research groups (Denver, CO and Rochester, NY) to assess the impact of centralized IIS-based influenza vaccine R/R, and to evaluate the effect of intensity of recall (1 v. 2 v. 3 reminders) over usual care. The investigators will also develop tools to aid other states in creating efficient IIS R/R systems for seasonal and possible pandemic influenza outbreaks.

This study has four aims.

Aim 1 is to develop the protocols, clinical decision support, and message content for state IISs to conduct reminder/recall for influenza vaccinations.

Aim 2 is to conduct a pragmatic trial, with randomization at the level of the patient within practices randomly selected to be proportionate to each state, to compare: 1) effectiveness and cost-effectiveness of centralized R/R of different intensity (1 vs. 2 vs. 3 messages) and usual care (0 messages) and 2) effectiveness and cost-effectiveness of R/R in specified subgroups (family medicine vs pediatric provider, rural vs urban, age of child) on receipt of influenza vaccination.

Aim 3 will measure the effect of adding mailed or text message R/R for autodialer failures vs. autodialer-alone R/R on influenza vaccination rates using a 2-arm Randomized Controlled Trial (RCT).

Aim 4 (dissemination aim) will develop a toolkit for state IIS-based influenza vaccine R/R for seasonal and pandemic influenza, and work with key stakeholders on a sustainability plan.

By the end of the study the investigators will have a feasible and cost-effective model to raise child seasonal or possibly pandemic influenza vaccination rates to prevent influenza. The investigators will disseminate the IIS model to all states.

ELIGIBILITY:
Inclusion Criteria:

* A record in the Colorado Immunization Information System,
* In need of at least one influenza vaccination at time of study,
* Affiliated with a participating practice, or
* Randomly selected among unaffiliated patients.

Exclusion Criteria:

* Opted out of participating in CIIS, or
* Are up-to-date on influenza vaccine

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56549 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects receiving influenza vaccine based on zero notices versus those receiving 1, 2 or 3 notices. | 6 months
  The primary outcome is receipt of influenza vaccine by children receiving zero notices compared to those receiving 1, 2 or 3 notices.

SECONDARY OUTCOMES:
Number of subjects receiving influenza vaccine based on demographic subgroups. | 6 months
  This outcome will categorize the number of influenza vaccines administered by subgroups, e.g.: Urban/Rural, Pediatrics/Family Practice, and age from 6m-1.9 yr., 2-10.9 yr. and 11-17.9 yr.
Number of subjects <9 years of age that will receive an additional vaccine. | 1 month
  If the subject is <9 years of age, they are required to received a second vaccine at least 1 month after receiving the initial vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Background] Kempe A, Saville AW, Dickinson LM, Beaty B, Eisert S, Gurfinkel D, Brewer S, Shull H, Herrero D, Herlihy R. Collaborative centralized reminder/recall notification to increase immunization rates among young children: a comparative effectiveness trial. JAMA Pediatr. 2015 Apr;169(4):365-73. doi: 10.1001/jamapediatrics.2014.3670. PMID 25706340
- [Result] Kempe A, Saville A, Dickinson LM, Eisert S, Reynolds J, Herrero D, Beaty B, Albright K, Dibert E, Koehler V, Lockhart S, Calonge N. Population-based versus practice-based recall for childhood immunizations: a randomized controlled comparative effectiveness trial. Am J Public Health. 2013 Jun;103(6):1116-23. doi: 10.2105/AJPH.2012.301035. Epub 2012 Dec 13. PMID 23237154
- [Derived] Kempe A, Saville AW, Albertin C, Helmkamp L, Zhou X, Vangela S, Dickinson LM, Tseng CH, Campbell JD, Whittington M, Gurfinkel D, Roth H, Hoefer D, Szilagyi P. Centralized Reminder/Recall to Increase Influenza Vaccination Rates: A Two-State Pragmatic Randomized Trial. Acad Pediatr. 2020 Apr;20(3):374-383. doi: 10.1016/j.acap.2019.10.015. Epub 2019 Nov 5. PMID 31698085